CLINICAL TRIAL: NCT05337189
Title: A Multicenter, Single-blind, Observational Clinical Trial of URISAFE
Brief Title: A Multicenter Clinical Trial of Urine DNA Testing for Bladder Cancer in China
Status: Recruiting | Type: Observational
Sponsor: Creative Biosciences (Guangzhou) Co., Ltd. (Industry)
Collaborators: Guangzhou Xiangkang Medical Research Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: KLM2021-04
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-06

CONDITIONS: Bladder Cancer; Urocystitis; Urinary Bladder Stone; Urothelial Carcinoma
Keywords: Bladder Cancer; Urine DNA Test; Gene Methylation Biomarkers; Multigene Methylation Detection; Cancer Screening; Urothelial Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Cystitis; Urinary Bladder Calculi; Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bladder cancer group: Two groups of sequential enrolled subjects, eligible subjects will be included in the study according to the inclusion criteria. In addition to collecting urine specimen for the testing kit of Human Multigene Methylation Detection Kit (Fluorescent PCR Method) test, eligible subjects also need to undergo the examination of standard method.
  Interventions: Diagnostic Test: Urine DNA methylation analysis; Procedure: medical imaging and/or cystoscopy and/or pathological examination
- The normal group: Two groups of sequential enrolled subjects, eligible subjects will be included in the study according to the inclusion criteria. In addition to collecting urine specimen for the testing kit of Human Multigene Methylation Detection Kit (Fluorescent PCR Method) test, eligible subjects also need to undergo the examination of standard method.
  Interventions: Diagnostic Test: Urine DNA methylation analysis; Procedure: medical imaging and/or cystoscopy and/or pathological examination

INTERVENTIONS:
Diagnostic Test: Urine DNA methylation analysis — Urine specimen will be collected by the subject for the detection of Human Multigene Methylation Detection Kit (Fluorescent PCR Method)
  Other Names: URISAFE
Procedure: medical imaging and/or cystoscopy and/or pathological examination — Subjects will undergo medical imaging and/or cystoscopy and/or pathological examination

SUMMARY:
The primary objective of this study is to assess the safety and effectiveness of Human Multigene Methylation Detection Kit (Fluorescent PCR Method) for help diagnose bladder cancer by comparing with clinical standard method (includes medical imaging (MRI, CT, etc.), cystoscopy, pathological examination).

DETAILED DESCRIPTION:
In this clinical trial, the testing kit to be evaluated is a Human Multigene Methylation Detection Kit (Fluorescent PCR Method), which is intended to qualitatively detect methylation levels of multiple genes in human urine specimen in vitro by Fluorescent PCR Method, and the standard method used in clinical diagnostic includes medical imaging, cystoscopy, pathological examination.

Subjects will provided urine specimen as required for the evaluation of the testing kit followed by a examination of standard method. Technical personnel who conduct the evaluation of the testing kit will remain blinded to the results of the clinical diagnosis.

The results of the testing kit will be compared with the standard method, and the effectiveness of the Human Multigene Methylation Detection Kit (Fluorescent PCR Method) for bladder cancer detection under normal clinical use will be assessed through statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject must meet all three of the following criteria to be eligible for the study:

  1. Who without age and gender limit, and is participating voluntarily and willing to sign Informed Consent Form;
  2. Who is willing to undergo or has completed medical imaging and/or cystoscopy and/or pathological examination;
  3. Any subject who is required to meet any of the following conditions:

     1. Who is diagnosed with or suspected of bladder cancer.
     2. Who has high risk factors for bladder cancer (such as engaged in contact with aromatic amines, dyes, rubber, aluminum, leather and other occupations, schistosomiasis infection, family genetic history, smoking, drinking, etc.).
     3. Who has hematuria symptoms (such as cystitis, stones, etc.).
     4. Who has other diseases that can be easily confused with bladder cancer.

Exclusion Criteria:

* Subject with any of the following conditions shall be excluded:

  1. Who has undergone surgery or chemoradiotherapy.
  2. Who has other conditions that the investigator considers inappropriate to participate in this clinical trial.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects without age limit, regardless of gender or region, and those who meet the inclusion criteria for this clinical trial, are eligible to enroll at the designated clinical sites. 482 subjects are targeted to enroll.
Sampling Method: Non-Probability Sample
Enrollment: 482 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | One year
  Sensitivity is the percentage of subjects with lung cancer who are correctly identified by the testing kit.
Specificity | One year
  Specificity is the percentage of subjects without lung cancer who are correctly excluded by the testing kit.
Consistency Rate | One year
  Consistency rate is the fraction of both true positive and negative diagnostic test results among all subjects.
Kappa Coefficient | One year
  Kappa coefficient is the consistency analysis of the extent of agreement between the test results of the testing kit and standard method.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Du, PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided
  We are carefully considering all applicable regulations and laws governing sharing of patients' data from China online with the global public.